CLINICAL TRIAL: NCT00884416
Title: Phase I Dose Finding Study of Sorafenib in Combination With Radiation Therapy and Temozolomide as a First Line Treatment of Patients With High Grade Glioma
Brief Title: Sorafenib in Newly Diagnosed High Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Andreas F. Hottinger, Principal Investigator, University Hospital, Geneva
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-122; 2009DR1029; 13031
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma
Keywords: high grade glioma; glioblastoma; gliosarcoma; anaplastic astrocytoma; anaplastic oligoastrocytoma; anaplastic oligodendroglioma; phase I; first line treatment; sorafenib; temozolomide; radiation therapy; safety; tolerability; protein kinase inhibitors
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib dose titration (Experimental)
  Interventions: Drug: Sorafenib dose escalation

INTERVENTIONS:
Drug: Sorafenib dose escalation — Sorafenib dose escalation scheme: 3 first patients: 200 mg/d, if dose limiting toxicities (DLT) not reached: 3 patients at 200 mg BID, if no DLT reached: 3 patients at 400 mg bid

SUMMARY:
This is a phase I study to evaluate the safety and tolerability of Sorafenib in combination with Temodar and radiation therapy in patients with newly diagnosed high grade glioma (glioblastoma, gliosarcoma, anaplastic astrocytoma and anaplastic oligodendroglioma or oligoastrocytoma). The mechanism of action of sorafenib, an oral multikinase inhibitor, makes it an interesting drug to investigate in the treatment of patients with high grade glioma as this agent has anti-angiogenic activity and inhibits other pathways such as Ras, Platelet-derived growth factor (PDGF) and fms-like tyrosine kinase receptor-3 (Flt-3), which are potential targets against gliomas.

DETAILED DESCRIPTION:
Up to 18 patients will be included in this phase I study. The primary goal of this study will be to establish the maximum tolerated dose of sorafenib when used in combination with temozolomide and radiation therapy. Secondary goals of this study include: response rate, time to treatment failure, 6 month progression-free survival, event free survival and overall survival. A correlative study will investigate the pharmacokinetics of sorafenib used in combination with radiation therapy and temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of newly diagnosed malignant glioma
* ECOG performance status of 0 or 1
* Age ≥18
* Life expectancy of at least 12 weeks
* Hemoglobin ≥ 9.0 g/dl
* Granulocyte count ≥1.5 X 10^9/L
* Platelet count ≥100 X 10^9/L
* SGOT ≤ 2.5X upper limit of normal (ULN)
* SGPT ≤ 2.5X upper limit of normal (ULN)
* Alkaline phosphatase ≤4x ULN
* Serum creatinine ≤1.5X ULN
* Bilirubin ≤1.5X ULN
* Spontaneous PT-INR/PTT < 1.5x upper limit of normal (patients on therapeutic anticoagulation will be allowed to participate.
* Patients must be on a stable or decreasing dose of corticosteroids for at least 2 weeks
* Patient for whom a first line treatment with temozolomide and radiotherapy is adequate
* Prophylactic anti-emetic, pentamidine inhalation / co-trimoxazole and anticonvulsants are allowed
* All patients must sign written informed consent.

Exclusion Criteria:

* Prior treatment for high grade glioma
* Previous exposure to Ras pathway inhibitors
* Other concurrent active malignancy (with the exception of cervical carcinoma in situ or non melanoma carcinoma of the skin, superficial bladder tumor [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry).
* Serious medical or psychiatric illness that would, in the opinion of the investigator, interfere with the prescribed treatment, including but not limited to: Congestive heart failure > NYHA class 2, active CAD, cardiac arrythmias requiring anti-arrythmic therapy or uncontrolled hypertension within the last 12 months
* Any condition limiting the patient's judgment capacity
* History of HIV infection, chronic hepatitis C or B as well as clinically active infections (> grade 2 NCI-CTC version 3.0)
* History of organ allograft
* Renal dialysis
* Evidence or history of bleeding diathesis
* Major surgery within 4 weeks of start of study treatment, except for neurosurgical resection
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.
* Medical condition that prevents the patient from swallowing pills
* Use of biologic response modifiers, such as G-CSF within 3 week of study entry.
* Pregnant or breast-feeding women.
* Refusal to use effective contraception. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and for at least 3 months after administration of study medication.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of sorafenib in combination with radiation and temozolomide chemotherapy | 35 weeks
  Safety and tolerability of sorafenib in combination with radiation and temozolomide chemotherapy in patients with newly diagnosed high grade glioma

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) and Area under the curve (AUC) of sorafenib and temozolomide | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post dose
Response rate | 35 weeks
Time to treatment failure | 20 months
6 month progression-free survival | 6 months
Event free survival | 20 months
Overall survival | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Dietrich, MD, Principal Investigator — Department of oncology, Geneva University hospital
Locations (1):
- Geneva University Hospital (Hopitaux Universitaires de Geneve), Department of Oncology, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Result] Hottinger AF, Ben Aissa A, Espeli V, Squiban D, Dunkel N, Vargas MI, Hundsberger T, Mach N, Schaller K, Weber DC, Bodmer A, Dietrich PY. Phase I study of sorafenib combined with radiation therapy and temozolomide as first-line treatment of high-grade glioma. Br J Cancer. 2014 May 27;110(11):2655-61. doi: 10.1038/bjc.2014.209. Epub 2014 May 1. PMID 24786603